CLINICAL TRIAL: NCT06244498
Title: Tranexamic Acid After Pathological Fracture Treated With Modular Arthroplasty: Retrospective Observational Study
Brief Title: Tranexamic Acid After Pathological Fracture Treated With Modular Arthroplasty
Status: Completed | Type: Observational
Sponsor: Piotr Biega (Other)
Responsible Party: Sponsor-Investigator, Piotr Biega, Principal Investigator, Rzeszow University of Technology - Assistant Professor, Podkarpackie Oncological Center
Organization: Podkarpackie Oncological Center (Other)
Other Study IDs: 01
Record Dates: First submitted 2024-01-12; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Metastases to Bone
Keywords: Blood Transfusion; Neoplasm Metastasis; Bone
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Tranexamic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TXA: Tranexamic acid was administered to the participants at a dose of 1.0 g during the induction of anaesthesia and immediately after the operation.
  Interventions: Drug: Tranexamic acid injection
- Non-TXA: Tranexamic acid were not administred to the participants .

INTERVENTIONS:
Drug: Tranexamic acid injection — Tranexamic acid were administered at a dose of 1.0 g during the induction of anaesthesia and immediately after surgery.
  Groups: TXA

SUMMARY:
This study assesses the safety and efficacy of TXA for patients treated for pathological femur fractures using modular prosthetics.

DETAILED DESCRIPTION:
Tranexamic acid is an efficacious medication for curtailing blood loss, haemoglobin drop, and the requirement for transfusions. Additionally, it is a secure medication, even when administered to oncology patients receiving reduction haemarthroplasty for pathological femoral fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patological fracture
* Arthroplasty using a modular prosthesis.

Exclusion Criteria:

* threatened fracture
* intraoperative blood transfusion
* fracture fixation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Investigetor analysed a group of paticipants who underwent surgery for metastatic tumours of the proximal femur using modular prostheses between 2017 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who require a blood transfusion. | During Hospitalization (up to day 10)
  Need of blood transfusion

SECONDARY OUTCOMES:
Estimeted blood lost after surgery. | During Hospitalization (up to day 3)
  Gross total blood loss was estimated utilizing the formula PBV × (Hctpre- Hctpost)/Hcta
Number of participants with embolic complication. | During Hospitalization (up to day 10)
  Yes or No

CONTACTS AND LOCATIONS:
Locations (1):
- SzSPOO Brzozów, Brzozów, Podkarpackie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analysed during the current study are available from the corresponding investigator on reasonable request.

REFERENCES:
- [Result] CRASH-2 collaborators; Roberts I, Shakur H, Afolabi A, Brohi K, Coats T, Dewan Y, Gando S, Guyatt G, Hunt BJ, Morales C, Perel P, Prieto-Merino D, Woolley T. The importance of early treatment with tranexamic acid in bleeding trauma patients: an exploratory analysis of the CRASH-2 randomised controlled trial. Lancet. 2011 Mar 26;377(9771):1096-101, 1101.e1-2. doi: 10.1016/S0140-6736(11)60278-X. PMID 21439633
- [Derived] Biega P, Guzik G. Tranexamic Acid Reduces Transfusion Rates After Modular Hemiarthroplasty for Pathological Femoral Fractures: A Retrospective Study. Adv Orthop. 2025 Oct 30;2025:3173784. doi: 10.1155/aort/3173784. eCollection 2025. PMID 41180854